CLINICAL TRIAL: NCT00472641
Title: Adjunctive Ziprasidone in Overweight and Obese Patients With Bipolar Disorder
Brief Title: Geodon in Weight Loss Study for Bipolar Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Terrence Ketter, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 96972
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ziprasidone/Geodon (Experimental): Ziprasidone/Geodon up to 320 mg per day
  Interventions: Drug: Ziprasidone/Geodon

INTERVENTIONS:
Drug: Ziprasidone/Geodon — Ziprasidone/Geodon

SUMMARY:
This research study is designed to determine if replacing your current antipsychotic and/or mood stabilizer with ziprasidone (Geodon) will impact weight. This research is being conducted because Geodon has a documented effect on mood. Additionally, we believe Geodon to be an effective medication for overweight or obese patients with bipolar disorder. There will be approximately 25 patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:Patients will meet the following criteria to be eligible to participate in the study:

* Diagnosis of Bipolar Disorder Type I, Type II, or NOS treated in ongoing therapy with atypical antipsychotic(s) and/or mood stabilizer(s) that have been implicated in causing weight gain (i.e. lithium, valproate, olanzapine, risperidone, quetiapine, aripiprazole).
* Age 18-65 years old
* Males; or nonpregnant, nonlactating females who are postmenopausal, surgically sterilized, or using a barrier method of contraception and have a negative pregnancy test
* Initial body mass index e 30 kg/m2, or e 27 kg/m2 and demonstrating or receiving treatment for metabolic consequences of overweight (fasting total cholesterol e 200mg/dL, fasting triglycerides e 250 mg/dL, or fasting blood glucose e 100 mg/dL).
* Stable medication regimen of at least one month
* Not have been hospitalized due to medical or psychiatric reasons during the past year from date of consent.
* Ability to understand and cooperate with study procedures
* Have signed a written informed consent prior to entering the study Exclusion Criteria:Patients may not participate in the study if they have any of the following conditions:
* One of the following DSM-IV Axis I diagnoses: delirium, dementia, amnestic and other cognitive disorders, schizophrenia, anorexia nervosa or bulimia, or substance abuse or dependence (active within the last month), abuse of illicit drugs (excluding marijuana) within the past month
* Antisocial personality disorder
* Medical complications of obesity such as diabetes, hypertension, hyperlipidemia, and cardiovascular disease unless followed by their own general medical practitioner who authorizes their participation in the trial, and continues to follow them medically and make necessary adjustments of concurrent antidiabetic, antihypertensive, antihyperlipidemic agents during the trial;
* Item 10 (Suicidal Thoughts) on the MADRS greater than or equal to 4
* Suicide attempt within the past three months
* Obesity of endocrine origin
* Seizure disorders
* Progressive neurologic or systemic disorders; HIV
* Other serious illnesses such as cardiac, hepatic (including cirrhosis), renal, respiratory, neurologic, or hematologic disease or glaucoma
* Hypothyroidism or hyperthyroidism unless adequately treated with TSH no more than 10% above or below the limits of the normal range.
* Administration of any investigational drug within 30 days prior to screening
* Allergy or hypersensitivity to ziprasidone
* Administration of clozapine in the prior three months
* Pregnancy within the past six months
* Patients will be discontinued from the study should they develop any significant adverse side effects that cannot be managed by dosage adjustment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Arthur Ketter, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Stanford University Bipolar Disorders Clinic — http://www.bipolar.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ziprasidone/Geodon
Started | 25
Completed | 18
Not Completed | 7
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone/Geodon
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Bipolar Subtype [Count of Participants; unit: Participants] — Bipolar I is characterized by one or more manic episodes or mixed episodes. Typically a person will experience periods of depression as well. Bipolar I disorder is marked by manic episodes. Bipolar II disorder is diagnosed after one or more major depressive episodes and at least one episode of hypomania, with possible periods of level mood between episodes.
  Bipolar disorder that does not follow a particular pattern is called bipolar disorder Not Otherwise Specified (NOS).
  Diagnosis follows criteria put forth by the DSM-4
  Participants
    Bipolar 1 | 10
    Bipolar 2 | 14
    Bipolar NOS | 1
Weight [Mean (Standard Deviation); unit: pounds] | 205.2 (31.7)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.9 (3.5)
Waist Circumference [Mean (Standard Deviation); unit: inches] | 41.7 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Was Weight Change From Baseline to Endpoint.
Description: The primary outcome measure will be the change in weight from baseline to endpoint using a random regression mixed effects model.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Ziprasidone/Geodon
Number analyzed (Participants) | 25
Pounds | -9.8 (7.5)
Statistical Analysis 1: Comparison: Ziprasidone/Geodon; Test type: Superiority or Other; p < 0.00001, Random Regression Mixed Effects Modeling

2. Secondary Outcome: Changes From Baseline to Endpoint in Body Mass Index (BMI)
Description: Secondary outcome measures will include the change from baseline to endpoint in Body Mass Index (BMI).
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Ziprasidone/Geodon
Number analyzed (Participants) | 25
kg/m^2 | 1.6 (1.2)
Statistical Analysis 1: Comparison: Ziprasidone/Geodon; Test type: Superiority or Other; p < 0.00001, Random Regression Mixed Effects Modeling

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Ziprasidone/Geodon
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone/Geodon (N=25)
Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Loss of Consciousness (Vascular disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypomania (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The current study has noteworthy limitations, including a small sample size, short trial duration, and an open, uncontrolled design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No